CLINICAL TRIAL: NCT04484597
Title: Predictors of COVID-19 Infection and Disease Progression
Acronym: Portsaiduni
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Other Study IDs: Prof. Refat Sadeq
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Positive COVID-19 by PCR
Keywords: COVID 19; Rt PCR; CT; Rapid tests
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rt PCR — positive COVID-19 by PCR and tested for other ancillary tests and CT chest to compare them and analyse which is the most sensitive in both moderate and severe clinical condition

SUMMARY:
Clinical Picture: Symptomatic COVID-19 presents with a recognizable clinical syndrome that is predictable prior to testing. Clinical judgement remains important, particularly when interpreting negative test results; 2. Biomarkers Associated with COVID-19 Patients: The most common laboratory features reported in patients with COVID-19

DETAILED DESCRIPTION:
The COVID-19 pandemic put tremendous pressures on the public health system and the health workers in almost every country around the world. Egypt was no exception, one of the main challenges faced is the limited number of CPR centers, equipment and kits which consequently affecting the number of tests that could be performed.

Although testing is critical, clinical judgement is the first mean to evaluate patients for COVID-19. Ancillary Diagnostic Tests and Chest imaging are also important tools before proceeding to the PCR testing. However, important gaps remain in screening asymptomatic persons in the incubation phase, as well as in the accurate determination of live viral shedding during convalescence to inform decisions to end isolation. The main objectives of the study: To set an evidence-based protocol with some criteria and procedures to reach - as accurate as possible - diagnosis without compromising the limited available resources. Such protocol shall make full use of the three main traditional pillars: Clinical picture, Ancillary Diagnostic Tests and Chest imaging before proceeding to the PCR testing:

1. Clinical Picture: Symptomatic COVID-19 presents with a recognizable clinical syndrome that is predictable prior to testing. Clinical judgement remains important, particularly when interpreting negative test results;
2. Biomarkers Associated with COVID-19 Patients: The most common laboratory features reported in patients with COVID-19 include: • Decreased albumin; • Elevated C-reactive protein ; • Elevated lactate dehydrogenase levels ; and • Lymphopenia .
3. Other biomarkers that have been reported include increased erythrocyte sedimentation rates; elevated aspartate aminotransferase, alanine aminotransferase, and creatine kinase levels, leukopenia, leukocytosis, increased bilirubin and creatinine levels. No biomarker or combination of biomarkers currently exists that is sensitive or specific enough to establish a diagnosis of COVID-19, or to pragmatically predict its clinical course.
4. Radiographic Tests: Many centers have evaluated the utility of chest imaging for diagnosis: • On chest radiography, bilateral pneumonia is the most frequently reported feature (range,11.8% to 100%) and is more common than a unilateral focus; • Computed tomography is regarded as more sensitive than radiography, with several cohort studies reporting that most patients (77.8% to 100%) had ground glass opacities. Other features commonly reported with COVID-19 on chest computed tomography include a peripheral distribution, fine reticular opacities, and vascular thickening. Compared with serial nasopharyngeal sampling, chest computed tomography may be more sensitive than an RT-PCR test at a single time point for the diagnosis of COVID-19. In addition, artificial intelligence may help distinguish COVID-19 from other etiologic agents of community-acquired pneumonia. However, these findings are not completely specific to COVID-19 and do not exclude a co-infection or an alternative diagnosis.

CPR: Who Should Be Tested? The current situation exemplifies the challenge of how to best utilize testing during outbreaks of novel pathogens. The initial testing criteria were too narrow to monitor and control the spread of the disease, but the sudden pivot to a far broader testing approach, even as capacity remains limited, may be an overcorrection. As of March 4, CDC discontinued specific guidance and recommends that "clinicians should use their judgment to determine if a patient has signs and symptoms compatible with COVID-19 and whether the patient should be tested," advising that "decisions on which patients receive testing should be based on the local epidemiology of COVID-19, as well as the clinical course of illness." High priorities for testing include patients with serious, unexplained respiratory illness and contacts of known cases, Methods: It is a comparative study between tests to diagnose COVID-19. In developed countries (in which Egypt is one of them) PCR is high cost. Though much of cases escape Diagnosis and clinician depend on clinical picture only. This study would allow to find what degree of dependence on other tests. In this study, 100 cases positive COVID-19 by PCR will be analyzed and tested for other ancillary tests and CT chest to compare them and find out which is the most sensitive in both moderate and severe clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* All cases positive COVID 19 RT PCR

Exclusion Criteria:

* cases with chronic diseases ( cancers, diabetes Liver or Kidney )

Min Age: 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: positive COVID-19 by PCR and tested for other ancillary tests and CT chest to compare them and analyse which is the most sensitive in both moderate and severe clinical condition
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
correlation of COVID-19 antibody to PCR | 1 year
  Finding the correlation between the results of COVID-19 RT PCR, antibody to PCR COVID-19 IgM & IgG and the severity of the clinical picture

SECONDARY OUTCOMES:
correlation of ancillaey tests to PCR | 1 year
  Finding the correlation between the results of the ancillary tests (CRP, ESR, LFT, Ferritin, D dimer) and the severity of the clinical picture

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Refat Sadeq, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: No